CLINICAL TRIAL: NCT02064127
Title: Evaluation of Triage Criteria for Abdominal Pain in the Emergency Department
Brief Title: Triage of Abdominal Pain in the Emergency Department
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Olivier T. Rutschmann, MD, MPH, University Hospital, Geneva
Other Study IDs: SU_2013_2
Record Dates: First submitted 2013-12-12; First posted 2014-02-17 (Estimated); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Abdominal Pain
MeSH Terms: conditions — Abdominal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with abdominal pain: Adult patients admitted to the Emergency Department with a main complaint of abdominal pain

SUMMARY:
The investigators aim to evaluate in a retrospective study the performance of the Swiss Emergency Triage Scale to identify at the door of the Emergency Department patients requiring emergent intervention.

DETAILED DESCRIPTION:
All patients are triaged at the door of our Emergency Department using the Swiss Emergency Triage Scale. Patients with abdominal pain may be triaged in two different emergency levels (level 2: medical evaluation within 20 minutes, level 3: medical evaluation within 2 hours). These levels are determined using a set of specific criteria.

The aim of this study is to evaluate the validity of these specific criteria in order to identify promptly patients with abdominal pain the will require an emergent intervention during their stay in the Emergency Department.

ELIGIBILITY:
Inclusion Criteria:

* >= 16 y
* abdominal pain as the main complaint

Exclusion Criteria:

* none

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults (> 16 y) admitted with abdominal pain in the Emergency Departement of a primary and tertiary teaching urban hospital.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Emergency intervention | participants will be followed for the duration of hospital stay, an expected average of 2 weeks
  Emergency intervention is a composite outcome of: emergency surgical intervention or radiological intervention or emergent endoscopy

SECONDARY OUTCOMES:
Time to medical evaluation | participants will be followed for the duration of emergency department stay, an expected average of 5 hours
  We will evaluate the delay between triage evaluation and medical evaluation. We will compute the percentage of patients evaluated within timeframe accordingly to the Swiss Triage Emergency Scale

CONTACTS AND LOCATIONS:
Overall Officials: Olivier T Rutschmann, MD, MPH, Principal Investigator — University Hospital, Geneva
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland